CLINICAL TRIAL: NCT04431076
Title: The PRO-PANC1 Project: Patient Reported Outcomes Measures to Predict Pancreatic Surgery Outcomes
Brief Title: Patient Reported Outcomes Measures to Predict Pancreatic Surgery Outcomes
Acronym: PRO-PANC1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massimo Falconi (Other)
Responsible Party: Sponsor-Investigator, Massimo Falconi, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: PRO-PANC1
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Patient Reported Outcome Measures; Quality of Life; Pancreatectomy; Nutritional Status; Recovery of Function
Keywords: Pancreatic cancer; Patient Reported Outcome Measures; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective single-center observational study with the mail objective to identify specific subgroups of patients planned for pancreatic resection, at high risk for postoperative morbidity and impaired recovery through preoperative screening of physical, functional, nutritional and psychological risk factors using patient reported questionnaires and performance tests.

Consecutive patients planned for pancreatic resection will be enrolled to screen for physical, functional, nutritional and psychological risk factors. The study duration is 3 years: 2 years of recruitment and 1 year of follow-up.

The findings of the present study will enable researchers to identify specific risk categories to plan personalized prehabilitation programs and modulate oncologic treatment strategies in cancer patients planned for pancreatic surgery.

DETAILED DESCRIPTION:
Patients undergoing pancreatic surgery, even treated in high-volume centers, still experience significant postoperative morbidity and full recovery after surgery takes longer than expected, delaying access to adjuvant oncologic treatment and influencing disease prognosis and patient quality of life. Patient health status at the time of surgery represents a major determinant of postoperative recovery. However, it is often evaluated with traditional measures such as performance status and comorbidity indices, which are frequently inaccurate and fail to capture the multiple dimensions of health and the patients' perspective.

Recent literature promotes the adoption of patient reported outcome measures (PROMs) to assess health across different domains (e.g. symptoms, functional status, well-being). These measures generally take the form of questionnaires and allow a more holistic understanding of patient's health and how surgery can affect different aspects of it. Thus, PROMs could be used as tools to identify patients at higher risk for postoperative adverse events or prolonged recovery.

Once higher risk profile patients have been identified, they could be referred to a for a personalized optimization program before surgery (i.e. prehabilitation). In fact, a few studies have recently enrolled high-risk patients candidate for major elective abdominal surgery in preoperative programs including multimodal interventions (e.g. physical activity, nutrition, mental exercise) resulting in decreased postoperative complications and earlier return of function. Optimizing preoperative status may reduce postoperative complications, enhance postoperative functional recovery and lead to shorter hospital stay, fewer readmissions, less time off work and improve patient perceived health-related quality of life.

Since high-risk patients benefit more from preoperative optimization strategies, and the implementation of a prehabilitation program is costly and resource-intensive, identifying patients at higher risk for postoperative poor outcomes is a key aspect. Unfortunately, there is no consensus on the best method to define these patients in the context of pancreatic surgery.

The main objective of this project is to identify specific subgroups of patients planned for pancreatic resection, at high risk for postoperative morbidity and impaired recovery through preoperative screening of physical, functional, nutritional and psychological risk factors using patient reported questionnaires and performance tests. The findings of the present study will enable researchers to identify specific risk categories to plan personalized prehabilitation programs and modulate oncologic treatment strategies in cancer patients planned for pancreatic surgery.

PRO-PANC1 is a prospective single-center observational study including consecutive patients planned for pancreatic resection to screen for physical, functional, nutritional and psychological risk factors.

Patients will be enrolled for 24 months and evaluated at the pre-admission visit (usually 1-2 weeks before surgery), at time of admission (i.e. the day before surgery), during hospital stay and trough a follow-up at 30 and 90 days, 6 and 12 monts after surgery. A navigator nurse who is already involved in patient follow-up after surgery will prompt patients to complete the questionnaires. There will be no additional visits or costs for patients and healthcare personnel in this activity.

PROMS (PATIENT REPORTED OUTCOMES MEASURES)

At their pre-admission visit, within 4 weeks before surgery, enrolled patients after signing the informed consent, will be asked to fill the following self-reported questionnaires:

* "Patient Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 (PROPr)", which is a flexible set of tools designed to measure self-reported physical, mental and social health and wellbeing which has been constructed and validated rigorously. It contains items from the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance and ability to participate in social roles and activities.
* Duke Activity Status Index (DASI) to evaluate patient physical status.
* Risk Analysis Index (RAI-C) to evaluate frailty, comorbidities and performance status.
* Patient Health Engagement scale (PHE-s) to assess patient engagement in their process of care based on their emotional and cognitive status.
* World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) - 12 items, a generic instrument to measure health and disability covering 6 domains of functioning.

PHYSICAL EVALUATION Physical performance testing will only be performed for a subgroup of patients in accordance with the availability of the physiotherapist and of the involved physician. Physical status will be evaluated by performace tests at the time of hospital admission (i.e. the day before surgery) for the baseline evaluation and at 30- days after surgery during the routine outpatient follow- up visit. The patient, either already admitted to the surgical ward, or during the outpatient evaluation will undergo testing with the physiotherapist in a dedicated area within the hospital (i.e. rehabilitation gym).

Performance tests will include: six-minute walk test, time up and go test, strength tests (target muscles will be the quadriceps and the handrip muscles: in both cases a specific dynamometer will be utilized) and the Modified Iowa Level of Assistance Scale (MILAS) evaluation.

In a subgroup of 100 cancer patients undergoing major pancreatic resection (pancreaticoduodenectomy and total pancreatectomy), preoperative cardiopulmonary exercise testing (CPET) will be administered. CPET is a non-invasive, dynamic test that provides a global assessment of the integrative responses to exercise.

NUTRITIONAL EVALUATION A baseline nutritional assessment will be performed at the pre-admission office visit or at the time of hospital admission (i.e. the day before surgery) by a study investigator. If the patient is already hospitalized, the evaluation will be performed at the patient bedside. The evaluation will include a nutrition history (e.g. weight loss, daily intake), measurement of anthropometric parameters including body weight (kg), height (cm), and body mass index (kg/m2). The Mini Nutritional Assessment (MNA) tool will be used to screen patients for nutrition risk. Standard biochemical markers of malnutrition and inflammation, including albumin, total proteins, total lymphocyte count, and C-reactive protein will be measured in all patients as part of the routine preoperative testing.

In a subgroup of patients, in accordance with the availability of the nutritionist, multi-frequency bioelectrical impedance vector analysis (BIVA) will be used to estimate total body water (TBW), extra-cellular water (ECW), fat free mass (FFM), fat mass (FM), body cell mass (BCM) and phase angle (PhA). This analysis will be performed at the time of the patient pre-admission visit or when the patient is admitted to the ward.

RADIOLOGIC EVALUATION Preoperative imaging (i.e. CT scan, MRI) performed within 30 days before surgery will be reviewed by a radiologist to evaluate pancreatic parenchyma morphological parameters with a potential impact on postoperative outcomes such as pancreatic duct size, pancreatic gland diameter, and fatty infiltration. Body composition parameters will also be evaluated including quantification of skeletal muscle area, visceral fat area, and subcutaneous fat area.

RISK SCORE ASSESSMENT Using a digital ecosystem platform, all information will be automatically captured and stored in the pancreatic disease institutional registry, in addition to other clinical information including laboratory tests, diagnostic imaging, pathology, and clinical history.

PROMS validity will be assessed in the context of pancreatic surgery according to the COSMIN recommendations for the design of the studiesy on measurement properties.

After evaluating the performance of each screening test, a practical risk scoring system for postoperative outcomes will then be developed based on regression models.

The newly developed score will then be released on a web page and app to allow researchers and clinicians to individually compute the score preoperatively to both inform patients of risks and to modify perioperative treatment strategies.

SAMPLE SIZE AND ANALYSIS The number of pancreatic resections at the San Raffaele Hospital Division of Pancreatic Surgery is around 330 per year. We assume that the rate of patients at high risk to develop postoperative complication is about 30%. Considering an overall rate of patients' refusal/not satisfying inclusion criteria/not performing physical or nutritional evaluation of 15%, we expect to enroll 561 patients in 24 months to have a hypothetical overall number of high risk patients of 168. After evaluating the performance of each screening test, a practical risk scoring system for postoperative outcomes will then be developed based on regression models.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age > 18 years) with pancreatic, biliary or duodenal diseases planned for pancreatic resection at San Raffaele Hospital
* Signed informed consent

Exclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) health status class 4-5.
* Patients with co-morbid medical, physical and mental conditions (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis), cardiac abnormalities, severe end-organ disease such as cardiac failure, morbid obesity (BMI >40), anemia (hematocrit < 30 %) and other conditions interfering with the ability to complete the performance testing procedures.
* Inability to read or understand Italian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients planned for pancreatic resection will be enrolled and screened for physical, functional, nutritional and psychological risk factors. The study duration is 3 years, patients will be recruited for 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Textbook outcome | 90 days after surgery
  Textbook outcome (TO) is a multidimensional measure for quality assurance, reflecting the "ideal" surgical outcome. TO is defined by the absence of clinically-relevant postoperative pancreatic fistula, bile leak, postpancreatectomy hemorrhage, severe complications (Clavien-Dindo ≥III) including mortality, and readmission.
  The primary outcome will be the failure to achieve a textbook outcome.
Postoperative complications | 90 days after surgery
  Postoperative complications occurring during the index admission or in a subsequent readmission, when related to surgery, will be recorded up to 90 days after surgery and graded by severity using the Dindo-Clavien classification and the Comprehensive Complication index (CCI).
  The Dindo-Clavien system grades complications according to the therapy needed for treatment: Grade I, are complications that require bedside management; Grade II, are complications that require pharmacologic treatment; Grade III, are complications that require surgical or radiologic intervention and; Grade IV, are complications that require intensive care treatment. Dindo-Clavien Grade III or above are considered severe postoperative complications.
  The CCI, derived from the Dindo-Clavien system, is a validated metric summarizing the complete spectrum of complications that occurred and their severity in a single score ranging from 0 to 100.
Pancreatic fistula | 90 days after surgery
  Occurrence of clinically-relevant postoperative pancreatic fistula defined as grade B or C POPF according to the 2016 International Study Group in Pancreatic Surgery (ISGPS) definition.

SECONDARY OUTCOMES:
Time to functional recovery | 90 days after surgery
  Time to functional recovery will be measured by subtracting the date of surgery from the date when participants achieve standardized criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self-care and no evidence of untreated medical problems).
Generic health related quality of life measured by Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile version 2.1 | 30 and 90 days after surgery
  Generic health-related quality of life will be measured using PROMIS-29+2, a questionnaire designed to measure self-reported physical, mental and social health status. It contains 29 questions covering seven domains of health. Questions are ranked on a 5-point Likert Scale. Each domain (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) is scored from 4 to 20. For negative domains (i.e. Depression), lower scores represent better outcomes, higher scores represent worse outcomes. For positive domains (i.e. Physical function), lower scores represent worse outcomes, higher scores represent better outcomes.
  Clinically meaningful minimally important differences for PROMIS scores are not established for our patient population. Difference in PROMIS scores for health domains between baseline and postoperative time points (30 and 90 days) will be considered to evaluate recovery after surgery.
Self reported physical activity - Duke Activity Status Index (DASI) | 30 and 90 days after surgery
  Self-reported activity status will be measured using the Duke Activity Status Index (DASI), a brief questionnaire designed to assess physical function and predict exercise capacity (peak oxygen uptake). Participants are asked to respond whether they are able to perform 12 listed activities of various intensities (ambulation, household tasks, personal care and leisure activities). A specific score is given for each positive answer. The possible total score range from 0 to 58. 0 corresponds to no activity (worse outcome); 58 corresponds to performance of all activities (best outcome).
Return to preoperative exercise capacity | 30 days after surgery
  This Secondary outcome includes the return at 30 days after surgery to preoperative exercise capacity as measured by the Six Minute Walk Test (6MWT).
  The 6MWT measures the total distance covered in 6 minutes of maximal walking effort.
  Patients will be considered to have recovered their exercise capacity when postoperative distance is within 20 meters of preoperative value or above.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò Pecorelli, Surgeon, Principal Investigator — Ospedale San Raffaele IRCCS
Locations (1):
- IRCCS San Raffaele, Milan, Italy